CLINICAL TRIAL: NCT02254967
Title: A Phase IIIB/IV Randomized, Controlled, Open-label, Parallel Group Study to Compare the Efficacy of Vancomycin Therapy to Extended Duration Fidaxomicin Therapy in the Sustained Clinical Cure of Clostridium Difficile Infection in an Older Population
Brief Title: A Phase IIIB/IV Study to Compare the Efficacy of Vancomycin Therapy to Extended Duration of Fidaxomicin Therapy in the Clinical Cure of Clostridium Difficile Infection (CDI) in an Older Population
Acronym: EXTEND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2819-MA-1002; 2013-004619-31 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Clostridium Difficile
Keywords: Aged; Fidaxomicin; Clostridium Difficile; Vancomycin
MeSH Terms: interventions — Fidaxomicin; OPT 80; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fidaxomicin Extended Pulsed Regimen (EPFX) (Experimental): Participants receive 200 mg fidaxomicin from day 1 to day 5 twice daily, followed by a 1-day gap (day 6) before starting alternate day dosing of 1 tablet of fidaxomicin 200 mg once daily from day 7 to day 25.
  Interventions: Drug: Fidaxomicin
- Vancomycin (Experimental): Participants receive 125 mg vancomycin from day 1 to day 10, 4 times daily.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin — oral tablets administered in an extended pulsed regimen
  Other Names: OPT-80; ASP2819; Dificlir; Dificid
  Arms: Fidaxomicin Extended Pulsed Regimen (EPFX)
Drug: Vancomycin — oral capsule
  Other Names: Vancocin
  Arms: Vancomycin

SUMMARY:
The main objective of the study is to evaluate whether the extended duration fidaxomicin therapy is superior to the standard vancomycin therapy in sustained clinical cure of CDI at 30 days after end of treatment (Day 40 or Day 55).

ELIGIBILITY:
Inclusion Criteria:

* CDI is confirmed by clinical symptoms (either > 3 unformed bowel movements or ≥ 200ml of unformed stool (for subjects having rectal collection devices)) in the 24 hours prior to randomization and CDI test confirmed positive for presence of C. difficile toxin A or B in stool within 48 hr prior to randomization.
* Subject agrees not to participate in another interventional study whilst participating in this study.

Exclusion Criteria:

* Subject is taking or requiring to be treated with prohibited medications
* Subject has received more than one day of dosing of any therapy for CDI within the last 48 hours
* Subject has experienced more than 2 previous episodes of CDI in the 3 months prior to study enrolment
* Subject is unable to swallow oral study medication.
* Subject has a current diagnosis of toxic megacolon.
* Subject is not willing to adhere to the provisions of treatment and observation specified in the protocol.
* Subject has been randomized into this study previously, has taken any investigational drug within 28 days or 5 half lives, whichever is longer, prior to enrollment, or is currently participating in another clinical study which may influence the assessment of efficacy and/or safety endpoints of this study, in the opinion of the Sponsor.
* Subject has previously participated in a CDI vaccine study
* Subject has hypersensitivity to fidaxomicin, vancomycin or any of its components.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-03-27 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Sustained Clinical Cure of CDI at 30 Days after End of Treatment | Day 40 (for vancomycin) and day 55 (for fidaxomicin extended pulsed regimen [EPFX])
  Sustained clinical cure is defined as an assessment of clinical response at test of cure (TOC; day 12 for vancomycin and day 27 or 12 for EPFX arm) and no recurrence of CDI from TOC until time of assessment. Clinical response is determined by the investigator based on the European Society of Clinical Microbiology and Infectious Diseases (ESCMID) criteria at TOC. Treatment response is present when either stool frequency decreases or stool consistency improves and parameters of disease severity (clinical, laboratory, radiological) improves and no new signs of severe disease develops.

SECONDARY OUTCOMES:
Percentage of Participants with a Sustained Clinical Cure of CDI at Day 40, Day 55 and Day 90 | Day 40, 55, 90
  Sustained clinical cure is defined as an assessment of clinical response at test of cure (TOC; day 12 for vancomycin and day 27 or 12 for EPFX arm) and no recurrence of CDI from TOC until time of assessment. Clinical response is determined by the investigator based on the ESCMID criteria at TOC. Treatment response is present when either stool frequency decreases or stool consistency improves and parameters of disease severity (clinical, laboratory, radiological) improves and no new signs of severe disease develops.
Percentage of Participants with a Clinical Response of CDI at 2 Days after End of Treatment | Day 12, 27
  Clinical response is determined by the investigator based on the ESCMID criteria (i.e., Treatment response is present when either stool frequency decreases or stool consistency improves and parameters of disease severity [clinical, laboratory, radiological] improves and no new signs of severe disease develops. Treatment response should be daily observed and evaluated after at least three days, assuming that the patient is not worsening on treatment) at TOC.
Percentage of Participants with a Clinical Response of CDI at Day 12 | Day 12
  Clinical response is determined by the investigator based on the ESCMID criteria (i.e., Treatment response is present when either stool frequency decreases or stool consistency improves and parameters of disease severity [clinical, laboratory, radiological] improves and no new signs of severe disease develops. Treatment response should be daily observed and evaluated after at least three days, assuming that the participant is not worsening on treatment) at TOC.
Number of Participants with a Relapse on Day 90 as Determined by Whole Genome Sequencing of C. Difficile Isolates | Baseline through day 90
  For participants with a recurrence after TOC, whole genome sequencing of isolates is performed on paired samples from day 1 and the day of the confirmed recurrence. Relapse is defined as paired isolates from a single recurrent participant with ≤ 2 single nucleotide variations (SNVs).
Time to Resolution of Diarrhea (TTROD) | Up to day 10 (for vancomycin) or up to day 25 (for EPFX)
  Time to resolution of diarrhea is defined as the time elapsing (in hours rounded up from minutes > 30) from the start of treatment (time of first dose of study drug) to resolution of diarrhea (time of the last unformed bowel movement [UBM] the day prior to the first of 2 consecutive days of ≤ 3 UBMs, > 50% reduction in number of stools or > 75% reduction in volume of liquid stool) that are sustained through to TOC.
Percentage of Participants with a Recurrence of CDI at Day 40, Day 55 and Day 90 | Day 40, 55, 90
  For participants with clinical response at TOC, recurrence of CDI is defined as re-establishment of diarrhea after TOC to an extent (judged by the frequency of passed UBMs) that is greater than the frequency recorded on day 10 for vancomycin arm or day 25 for EPFX arm (2 days prior to TOC), confirmed by a CDI test positive for Toxin A/B and requiring further CDI therapy.
Time to Recurrence of CDI after End of Active Treatment | From day 10 up to day 90
  Time to recurrence of CDI is defined as the time in days from clinical response until onset of recurrence of CDI for participants who respond at TOC.
Disease-free Survival After Day 10 | From day 10 up to day 90
  Disease-free survival is defined as the time in days a participant does not have symptoms of diarrhea from day 10 up to day 90 for participants who respond at TOC.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe Ltd.
Locations (109):
- Austria (3):
  - Site AT43002, Graz
  - Site AT43003, Linz
  - Site AT43001, Salzburg
- Belgium (5):
  - Site BE32007, Aalst
  - Site BE32006, Bruges
  - Site BE32001, Brussels
  - Site BE32005, Brussels
  - Site BE32008, Liège
- Croatia (4):
  - Site HR38506, Osijek
  - Site HR38503, Rijeka
  - Site HR38505, Zadar
  - Site HR38501, Zagreb
- Czechia (5):
  - Site CZ42002, Brno-Bohunice
  - Site CZ42005, Kyjov
  - Site CZ42004, Opava
  - Site CZ42003, Prague
  - Site CZ42001, Praha 8 - Libeň
- Denmark (3):
  - Site DK45001, Herlev
  - Site DK45005, Hillerød
  - Site DK45004, Nykøbing Falster
- Finland (2):
  - Site FI35801, Helsinki
  - Site FI35802, Turku
- France (9):
  - Site FR33003, Bordeaux
  - Site FR33008, Clermont-Ferrand
  - Site FR33006, Lille
  - Site FR33005, Nantes
  - Site FR33004, Nîmes
  - Site FR33001, Paris
  - Site FR33007, Paris
  - Site FR33002, Rennes
  - Site FR33009, Saint-Priest-en-Jarez
- Germany (6):
  - Site DE49001, Cologne
  - Site DE49011, Cologne
  - Site DE49012, Hamburg
  - Site DE49006, Leipzig
  - Site DE49016, Lübeck
  - Site DE49008, Marburg
- Greece (9):
  - Site GR30005, Athens
  - Site GR30008, Athens
  - Site GR30001, Athens
  - Site GR30004, Athens
  - Site GR30009, Athens
  - Site GR30007, Athens
  - Site GR30002, Herakleion, Crete
  - Site GR30006, Larissa
  - Site GR30010, Thessaloniki
- Hungary (8):
  - Site HU36004, Békéscsaba
  - Site HU36010, Budapest
  - Site HU36009, Budapest
  - Site HU36001, Debrecen
  - Site HU36006, Gyula
  - Site HU36005, Mosonmagyaróvár
  - Site HU36008, Orosháza
  - Site HU36007, Pécs
- Ireland (2):
  - Site IE35302, Dublin
  - Site IE35304, Limerick
- Italy (9):
  - Site IT39009, Florence
  - Site IT39005, Genova
  - Site IT39004, Milan
  - Site IT39003, Monza
  - Site IT39007, Napoli
  - Site IT39002, Padua
  - Site IT39001, Pisa
  - Site IT39006, Roma
  - Site IT39010, Torino
- Poland (6):
  - Site PL48012, Lodz, PL
  - Site PL48004, Gdynia
  - Site PL48011, Szczecin
  - Site PL48008, Warsaw
  - Site PL48002, Warsaw
  - Site PL48003, Zgierz
- Portugal (5):
  - Site PT35101, Almada
  - Site PT35102, Amadora
  - Site PT35106, Cotter
  - Site PT35104, Vila Nova de Gaia
  - Site PT35107, Vila Real
- Romania (3):
  - Site RO40001, Bucharest
  - Site RO40003, Cluj-Napoca
  - Site RO40002, Lasi
- Russia (2):
  - Site RU70001, Moscow
  - Site RU70003, Moscow
- Slovenia (4):
  - Site SI38601, Ljubljana
  - Site SI38605, Ljubljana
  - Site SI38602, Maribor
  - Site SI38603, Murska Sobota
- Spain (4):
  - Site ES34003, Barakaldo, Vizcaya
  - Site ES34004, Barcelona
  - Site ES34005, Madrid
  - Site ES34006, Valencia
- Sweden (4):
  - Site SE46002, Gothenburg
  - Site SE46004, Jönköping
  - Site SE46001, Lund
  - Site SE46005, Uppsala
- Switzerland (3):
  - Site CH41001, Lugano, Canton Ticino
  - Site CH41002, Sankt Gallen
  - Site CH41004, Zurich
- Turkey (Türkiye) (7):
  - Site TR90003, Adana
  - Site TR90002, Ankara
  - Site TR90007, Ankara
  - Site TR90001, Antalya
  - Site TR90006, Eskişehir
  - Site TR90005, Istanbul
  - Site TR90004, Istanbul
- United Kingdom (6):
  - Site GB44003, Sutton in Ashfield, Nottinghamshire
  - Site GB44006, Bristol, UK
  - Site GB44008, Blackpool
  - Site GB44005, Cardiff
  - Site GB44010, London
  - Site GB44009, Truro

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Cornely OA, Vehreschild MJGT, Adomakoh N, Georgopali A, Karas A, Kazeem G, Guery B. Extended-pulsed fidaxomicin versus vancomycin for Clostridium difficile infection: EXTEND study subgroup analyses. Eur J Clin Microbiol Infect Dis. 2019 Jun;38(6):1187-1194. doi: 10.1007/s10096-019-03525-y. Epub 2019 Mar 25. PMID 30911926
- [Derived] Guery B, Menichetti F, Anttila VJ, Adomakoh N, Aguado JM, Bisnauthsing K, Georgopali A, Goldenberg SD, Karas A, Kazeem G, Longshaw C, Palacios-Fabrega JA, Cornely OA, Vehreschild MJGT; EXTEND Clinical Study Group. Extended-pulsed fidaxomicin versus vancomycin for Clostridium difficile infection in patients 60 years and older (EXTEND): a randomised, controlled, open-label, phase 3b/4 trial. Lancet Infect Dis. 2018 Mar;18(3):296-307. doi: 10.1016/S1473-3099(17)30751-X. Epub 2017 Dec 19. PMID 29273269
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;2819-MA-1002